CLINICAL TRIAL: NCT06694870
Title: Transcutaneous CO2 Measurement - From Hospital to Home
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marte Skogstad Allgot, Cand.med, University of Oslo
Other Study IDs: 707967
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Respiratory Failure; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Hypoventilation; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital: Transcutaneous monitoring in the hospital
  Interventions: Diagnostic Test: Transcutaneous CO2 monitoring
- Home: Transcutaneous monitoring at home
  Interventions: Diagnostic Test: Transcutaneous CO2 monitoring

INTERVENTIONS:
Diagnostic Test: Transcutaneous CO2 monitoring — Transuctaneous CO2 monitoring

SUMMARY:
Long-term non-invasive ventilation (LT-NIV) is the main treatment modality for chronic hypercapnic respiratory failure.To assess the adequacy of alveolar ventilation during sleep and potential sleep hypoventilation, nocturnal transcutaneous CO2 (PtcCO2) monitoring is necessary. There is an increased tendency to monitor patients at home, but there is a lack of robust data comparing the technical success rates between the home and inpatient setting of PtcCO2 monitoring. The primary aim of the current study was to evaluate the rate of successful nocturnal PtcCO2 monitoring in a home setting in a population of patients with chronic hypercapnic respiratory failure receiving LT-NIV. The secondary aim was to compare these data with PtcCO2 registrations performed during regular follow up of a similar population of patients in a hospital setting.

DETAILED DESCRIPTION:
Patients scheduled for LT-NIV follow-up at Oslo University Hospital, Ullevål in the time-period January 2020 to December 2022 were prospectively identified. Follow-up monitoring occurred either at home or in the hospital. Two physicians blinded to the location of the monitoring, retrospectively classified the PtcCO2 as successful or unsuccessful, and identified the causes of failure for the latter.

ELIGIBILITY:
Inclusion criteria for both groups were:

1. LT-NIV treatment for at least 3 months,
2. that the monitoring was due to a scheduled follow-up appointment,
3. at least one follow-up visit at the hospital after LT-NIV initiation. Inclusion in the study required a signed consent from all participants.

There were three additional criteria for the home monitoring group:

1. home address in reasonable proximity to the hospital,
2. the subject/spouse/assistant/home health care provider was assumed capable of operating the equipment, and
3. the subject consented to undertaking the monitoring at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Demographics Total Subjects (n) 129 Male 76 (59.0%) Age (mean) 54,9 ±18.0 Diagnosis Neuromuscular disorders: 85 (65.9%) COPD 9 (7.0%) Obesity hypoventilation syndrome: 24 (18.6%) Restrictive: 11 (8.5%)
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Success rate home vs hospital | January 1st 2020 - December 31st 2022

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Aarrestad, Dr.med, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No